CLINICAL TRIAL: NCT03487029
Title: The Effects of Different High-intensity Interval Training Training Protocols on Cardiorespiratory Parameters in Patients With Type 2 Diabetes
Brief Title: High-intensity Interval Training Training Protocols on Cardiorespiratory Parameters in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cemile Bozdemir Ozel, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA17069
Record Dates: First submitted 2018-02-06; First posted 2018-04-03 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Diabetes
Keywords: diabetes; high intensity interval training; cardiorespiratory fitness
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short duration group (Experimental): 30sn %100 Wmax 120sn %25 Wmax 3 sessions/week total 8 weeks
  Interventions: Other: Short duration
- long duration group (Experimental): 4dk %85 Wmax 120sn %25 Wmax 3 sessions/week total 8 weeks
  Interventions: Other: Long duration

INTERVENTIONS:
Other: Short duration — exercise Short duration high intensity training
  Other Names: training
  Arms: short duration group
Other: Long duration — exercise Long duration high intensity training
  Other Names: training
  Arms: long duration group

SUMMARY:
Aim: To assess whether there are different training effects on glucose concentration and cardiorespiratory parameters of different high-intensity training protocols in patients with type 2 diabetes.

Type 2 diabetes is a highly prevalent disease associated with cardiovascular disease leading to high levels of mortality, morbidity and health expenditure, characterized by impaired glucose control during activities and reduced aerobic exercise capacity .

Exercise training is the most effective way to improve compliance, reduce blood glucose concentration and increase insulin sensitivity. Training increases muscle capacity, oxidative capacity and glucose transport, peripheral insulin sensitivity is improved.

Exercise training with high-intensity interval (resting and exercise period) High Intensity Interval Training (HIIT) is a form of exercise training that has recently been widely used in the management of type 2 diabetes, including short duration high intensity exercise periods and lower severity or passive rest periods. There are different HIIT exercise training programs according to physiological responses in the literature. However, long-term and short-term HIIT training training programs were not compared in terms of their effect on glucose concentration and cardiorespiratory fitness. The aim of this study was to compare the effects of different HIIT exercise training programs so that exercise programs for patients with type 2 diabetes could be planned more effectively.

DETAILED DESCRIPTION:
This study will be participated patients with Type 2 diabetes. Patients' laboratory values, pulmonary function test, respiratory muscle strength, exercise capacity, physical activity level, quality of life will be evaluated.

Pulmonary function test will be assesed with spirometer, respiratory muscle strength will be evaluated with mouth pressure. Exercise capacity will be evaluated using six minute walking test, incremental shuttle walk test, cycle ergometer. Muscle oxigeneration will be asssed with wearable lactate threshold predicting device. Physical activity level will be evaluated trial accelerometer.

Then, patients will be randomly divided two high intensity interval exercise training groups.

First group: short duration high intensity exercise training (Exercise load phase : 30sn %100 Patients performance, rest phase: 120sn %25 patients performance) Second group: Long duration high intensity interval exercise training (Exercise load phase : 4 dk %100 Patients performance, rest phase: 120sn %25 patients performance) All patients will participate three times a week during eight weeks. The muscle oxigeneration, blood glucose consantration, blood pressure, heart rate will be recorded before and after each exercise session. After 8 week, all test will be done again.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes
* aged 18-64 years
* patients can walk and cooperative
* body mass index is less than 40 kg / m2

Exclusion Criteria:

Individuals have known lung disease,have undergone any cardiac event or surgery within the past six months, have uncontrolled hypertension, and have diabetic complications such as nephropathy, retinopathy and severe neuropathy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
muscle oxigeneration | Change from baseline muscle oxigeneration at 8 weeks
  It is evaluate with wearable lactate threshold device on gastrocinemius

SECONDARY OUTCOMES:
The blood glucose consentration | before and after 8 weeks
  It is evaluate with sample from blood
Functional Exercise capacity | before and after 8 weeks
  İt is evaluated with six minute walk test
Maximal exercise capacity | before and after 8 weeks
  İt is evaluated using with incremental shuttle test
Symptom limited maximal exercise capacity | before and after 8 weeks
  İt is evaluated with cycle ergometer test
Lipit profile-High density lipoprotein cholesterol | before and after 8 weeks
  High density lipoprotein cholesterol wiil be assesed
Lipit profile- low density lipoprotein cholesterol | before and after 8 weeks
  low density lipoprotein cholesterol wiil be assesed
Lipit profile- trigliseride | before and after 8 weeks
  trigliseride wiil be assesed
pulmonary parameter-Forced vital capacity | before and after 8 weeks
  Forced vital capacity will be evaluated
pulmonary parameter-Forced vital capacity in the first second | before and after 8 weeks
  Forced vital capacity in the first second will be evaluated
pulmonary parameter-Mid expiratory flow rate | before and after 8 weeks
  Mid expiratory flow rate will be evaluated
pulmonary parameter-Peak expiratory flow | before and after 8 weeks
  Peak expiratory flow will be evaluated
Respiratory muscle strength | before and after 8 weeks
  It is evaluated with mouth pressure
Physical activity level | before and after 8 weeks
  ıt is assessed using accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Bozdemir Özel, McS, Principal Investigator — Hacettepe University Physiotherapy and Rehabilitation
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)